CLINICAL TRIAL: NCT03543878
Title: Stimulating Neural Activity to Improve Blood Flow and Reduce Amyloid: Path to Clinical Trials
Acronym: FLICKER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, James Lah, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB00101694
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Flicker Fusion

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two study arms. One group will receive the Flicker exposure for 8 weeks while the other group will receive the active exposure for 4 weeks.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Flicker for 8 Weeks (Experimental): Participants will receive the Flicker exposure during the entire 8-week treatment period
  Interventions: Device: Flicker
- Flicker for 4 Weeks (Active Comparator): Participants will receive the Flicker exposure during the second four weeks of the 8-week treatment period
  Interventions: Device: Flicker

INTERVENTIONS:
Device: Flicker — The Flicker intervention is delivered with the GammaSense Stimulation System by Cognito Therapeutics and involves viewing flickering lights at gamma frequency (like a strobe light but faster) to drive gamma oscillations in visual brain areas. The GammaSense Stimulation System is a device consisting of a pair of opaque glasses with a light-emitting diode (LED) illumination on the interior of the glasses. Headphones worn by the user during the stimulation session provide the auditory stimulation. When activated for the treatment session, the device will generate light and sound oscillations at 40 cycles per second (Hz) for 60 minutes. Participants will use the device daily during their active treatment period.
  Other Names: driving gamma; GammaSense Stimulation System

SUMMARY:
Alzheimer's disease is characterized by the accumulation of toxic proteins in the brain. Mechanisms to remove these proteins have been the target of many drug trials. This study is designed to use a device to entrain brain waves to a specific frequency to see if rodent research can be replicated in humans with mild cognitive impairment. Ten participants will be recruited from the Emory Alzheimer's Disease Research Center (ADRC) database and assigned to either treatment for 8 weeks or treatment for 4 weeks. This latter group will serve as the control group (4 weeks no treatment, 4 weeks treatment). It is hypothesized that exposure to the gamma oscillations (Flicker) will clear toxic proteins from the brain and increase cerebral blood flow.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is a looming epidemic, with an urgent need for new therapies to delay or prevent symptom onset and progression. There is growing awareness that clinical trials must target stage-appropriate pathophysiological mechanisms to effectively develop disease-modifying treatments. Advances in AD biomarker research have demonstrated changes in amyloid, brain metabolism, and other pathophysiologies prior to the onset of memory loss, with some markers possibly changing one or two decades earlier. The brain region responsible for spatial navigation and memories of experience, the hippocampus, is one of the areas first affected in Alzheimer's disease (AD) and other memory disorders. Prior research has shown how coordinated electrical activity across many neurons in the hippocampus represents memories of experiences and this coordinated activity fails in animal models of AD. The research also showed that stimulating neurons to produce a specific component of this activity, called gamma oscillations, reduces AD pathology. The goal of this proposal is to translate this discovery that stimulating specific patterns of neural activity is neuroprotective from rodents to humans using a non-invasive approach. This research includes preclinical testing that will be used to design and justify a multi-site clinical trial to test this approach as a treatment for AD, for which there are currently no effective therapies.

Cognito Therapeutics has licensed the technology from prior animal research to transition this work to humans. The company will provide the Flicker devices for conducting this study. The device is similar to sunglasses and is both comfortable and easy to use.

Ten participants with mild cognitive impairment will be randomly assigned to two study arms. Although all participants will receive Flicker exposure, half of the participants will receive the exposure during the entire intervention period (8 weeks of Flicker) while the other half of the participants will receive Flicker exposure only during the second half of the intervention period (for 4 weeks of active treatment). During the course of the study, participants will undergo venous blood draws and lumbar puncture for biomarker analyses at baseline, midpoint and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a subjective memory concern as reported by subject, study partner or clinician.
* Meets local criteria for diagnosis of mild cognitive impairment (MCI).
* Montreal Cognitive Assessment (MoCA) score >15. Exceptions may be made for subjects with less than 8 years of education at the discretion of the PI.
* Clinical Dementia Rating = 0.5. Memory Box score must be at least 0.5.
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's Disease (AD) cannot be made by the physician at the time of the screening visit.
* Stable on medications for 4 weeks prior to initiation of study sessions.
* Geriatric Depression Scale (GDS) ≤ than 6.
* Male or female outpatients aged 50-90 (inclusive).
* Able to hear without the use of hearing aids.
* Study partner who lives with the participant and can provide a reliable assessment of the participant's level of function, is available for all clinic visits, and can serve as a supervisor/monitor for the home-based Flicker sessions for the duration of the study.
* Visual and auditory acuity adequate for neuropsychological testing.
* Good general health with no diseases expected to interfere with the study.
* Completed six grades of education or has a good work history (sufficient to exclude mental retardation).
* Able to communicate in English with study personnel.
* Able to understand the nature of the study and provision of written informed consent prior to conduct of any study procedures.
* Willing to undergo repeated magnetic resonance imaging (MRI) and positron emission tomography (PET) scans.
* Agrees to blood collection for apolipoprotein E (ApoE) and biomarker testing.
* Agrees to lumbar puncture over the course of the study for the collection of cerebrospinal fluid (CSF).

Exclusion Criteria:

* Any significant neurologic disease other than MCI and suspected incipient AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, poorly controlled seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic deficits or known structural brain abnormalities.
* Screening/baseline MRI scan with evidence of infection, large vessel infarction or other focal structural lesions that could account for the memory deficits. Subjects with multiple lacunes or lacunes in a critical memory structure are excluded.
* Contraindication to MRI due to pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments or foreign objects in the eyes, skin or body, or excessive weight.
* Presence of clinically significant suicide risk, based on the Investigator's judgment informed by a structured clinician interview. Any suicide attempt within the past 1 year of the screening visit is exclusionary.
* Major depression, bipolar disorder as described in Diagnostic and Statistical Manual of Mental Disorders-4 (DSM-IV) within the past 1 year, or history of schizophrenia.
* Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM-IV criteria).
* Known history of epilepsy or migraines, which may be exacerbated by study intervention.
* History of narrow angle (acute angle) glaucoma.
* Current use of warfarin or other blood thinners (exclusionary for lumbar puncture).
* Inability to obtain initial CSF sample.
* Current use of Namenda (memantine).
* Current use of medications that lower seizure threshold, including Wellbutrin, Ciprofloxacin, Levofloxacin, Seroquel, Phenergan, and Sumatriptan.
* Current use of anti-psychotic medication.
* CSF profile inconsistent with underlying Alzheimer's Disease pathology.
* Reasonable likelihood for non-compliance with the protocol or any other reason, in the opinion of the investigator, prohibits enrollment of subject into the study.
* Exceptions to these guidelines may be considered on a case-by-case basis at the discretion of the protocol director.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-11-16 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Lah, MD, PhD, Principal Investigator — Emory University
Locations (1):
- 12 Executive Park Drive, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Emory Cognitive Neurology Clinic and the Emory Goizueta Alzheimer's Disease Research Center (ADRC), in Atlanta, Georgia. Participant enrollment began on November 16, 2018 and study follow up was completed on February 10, 2020.
Groups:
- Flicker/Flicker: Participants receiving the Flicker exposure for the first 4 weeks of the study and the second four weeks of the study, for a total of 8 weeks of treatment.
- No Flicker/Flicker: Participants receiving no exposure to Flicker for the first 4 weeks of the study and then receiving the Flicker exposure for the second four weeks of the study, for a total of 4 weeks of treatment.
Period: Overall Study
Arm/Group | Flicker/Flicker | No Flicker/Flicker
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flicker/Flicker | No Flicker/Flicker | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 72 (8.15) | 70.6 (6.54) | 71.3 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 2 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Adherence to Daily Device Use
Description: Feasibility of the Flicker intervention is defined as adherence to Flicker exposure, at home, for one hour per day for the duration of the intervention period (4 or 8 weeks). The percentages of completed sessions are presented here.
Time Frame: Week 8
Measure: Mean (Standard Deviation); unit: percentage of adherence to treatment
Arm/Group | Flicker/Flicker | No Flicker/Flicker
Number analyzed (Participants) | 5 | 5
percentage of adherence to treatment | 95.55 (2.92) | 95.37 (4.72)

2. Primary Outcome: Percentage of Maximum Tolerated Stimulation
Description: Participants rated their tolerance to Flicker stimulation prior to the study intervention, using a 1 - 5 point Likert scale for each of the 10 levels of brightness (visual stimulation) and each of the 10 levels of loudness (auditory stimulation) after 60 seconds of stimulation at each level. A rating of 1 indicated stimulation "can be withstood and comfortable," 3 indicated stimulation is "tolerable, but not necessarily comfortable," and 5 indicated stimulation "cannot be withstood or is uncomfortable." Ratings of 1, 2, and 3 were considered tolerable. After determining tolerance for auditory and visual stimulation separately, participants were exposed to combined visual and auditory levels beginning one level above the participant's highest stimulation that received a rating of 3 or lower. Tolerability of brightness and loudness levels of combined auditory stimulation was assessed for 60 seconds. See Analysis Population Description for more details.
Time Frame: Baseline
Population: Outcome Measure Description continued: Tolerability at the highest level of "10" was scored as 100. Maximum tolerated levels for visual alone, auditory alone, visual combined, and auditory combined were averaged for the Flicker/Flicker and No Flicker/Flicker groups.
Measure: Mean (Standard Deviation); unit: percentage of tolerated stimulation
Groups:
- All Study Participants: Participants receiving the Flicker exposure in either the Flicker/Flicker or No Flicker/Flicker study arm.
Arm/Group | All Study Participants
Number analyzed (Participants) | 10
percentage of tolerated stimulation
  Visual alone | 94 (9.66)
  Auditory alone | 98 (4.22)
  Visual when combined with auditory | 93 (12.52)
  Auditory when combined with visual | 94 (18.97)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the time when participants were receiving the Flicker intervention (up until Week 8 for the Flicker/Flicker group and until Week 4 for the No Flicker/Flicker group).
Arm/Group | Flicker/Flicker | No Flicker/Flicker
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 4/5 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flicker/Flicker (N=5) | No Flicker/Flicker (N=5)
Dizziness (General disorders) | 0 | 1 — possibly related to study treatment
Tinnitus (Ear and labyrinth disorders) | 1 | 0 — possibly related to study treatment
Headache (General disorders) | 1 | 0 — possibly related to study treatment
Double vision (General disorders) | 0 | 1 — not related to study treatment
Leg, arm, joint pain (Musculoskeletal and connective tissue disorders) | 1 | 1 — not related to study treatment
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 — not related to study treatment
Depression (Psychiatric disorders) | 1 | 0 — not related to study treatment
Rhinorrhea (General disorders) | 1 | 0 — not related to study treatment
Gastrointestinal problems (General disorders) | 1 | 0 — not related to study treatment
Fall (Injury, poisoning and procedural complications) | 0 | 1 — not related to study treatment
Dog bite (Injury, poisoning and procedural complications) | 0 | 1 — not related to study treatment
Skin growth on neck (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 — not related to study treatment
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 — not related to study treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/78/NCT03543878/Prot_SAP_000.pdf